CLINICAL TRIAL: NCT01874860
Title: Preemptive Therapy Study of Cetuximab(Erbitux®)Induced Skin Rash Using Doxycycline, Sunscreen, Hydrocortisone and Moisturizer in Colorectal and Head and Neck Cancer Patients
Brief Title: Skin Rash Study Before Chemotherapy in Colorectal & Head and Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Rebecca Redman, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCC-OHN-GI-13
Record Dates: First submitted 2013-06-06; First posted 2013-06-11 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer; Head and Neck Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms | interventions — Doxycycline; Hydrocortisone; Sunscreening Agents; Clindamycin; Gels; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extensive treatment group (Experimental): Doxycycline capsule, 100 mg, taken twice daily; sunscreen SPF 30 or higher applied to exposed skin areas at least 30 minutes before going outdoors each morning; moisturizer applied to the face, hands, feet, neck, back, and chest each morning after sunscreen; Hydrocortisone 1% topical cream applied to the face, hands, feet, neck, back, and chest each evening.
  For patients with grade 1 rash, hydrocortisone 1% cream and clindamycin 1% gel (tetracycline antibiotic) are recommended for daily use.
  For patients with grade 2 rash, hydrocortisone cream and doxycycline 100mg twice daily or minocycline (tetracycline antibiotic) 100mg once daily is recommended.
  For patients with grade 3 rash, systemic steroid therapy (a Medrol dose-pack) will be added to the grade 2 treatment.
  Interventions: Drug: Doxycycline; Drug: Hydrocortisone 1% cream; Other: Sunscreen; Other: Moisturizer; Drug: Clindamycin; Drug: Medrol-dose pack (Steroid)
- Standard care group (Experimental): Patient will not receive preventive treatment but will be allowed to use sunscreen and moisturizer if desired.
  Interventions: Other: Sunscreen; Other: Moisturizer

INTERVENTIONS:
Drug: Doxycycline — Doxycycline capsule, 100 mg, taken twice daily
  Arms: Extensive treatment group
Drug: Hydrocortisone 1% cream — Applied to the face, hands, feet, neck, back, and chest each evening (Topical cream)
  Arms: Extensive treatment group
Other: Sunscreen — Applied to exposed skin areas at least 30 minutes before going outdoors each morning.
  Other Names: SPF 30 or higher sunscreen
Other: Moisturizer — Applied to the face, hands, feet, neck, back, and chest each morning after sunscreen
  Other Names: Any frangrance-free moisturizer will do
Drug: Clindamycin — Recommended for daily use if rash returns (Topical cream)
  Other Names: Clindamycin 1 % gel
  Arms: Extensive treatment group
Drug: Medrol-dose pack (Steroid) — Patients will receive a Medrol dose-pack while continuing the extensive treatment regimen.
  Other Names: Medrol-dose pack
  Arms: Extensive treatment group

SUMMARY:
The purpose of this study is to determine if using preventive treatments such as Doxycycline (an anti-biotic) capsules, sunscreen with SPF 30, Hydrocortisone 1% cream and a moisturizer will help to reduce the incidence and severity of the skin rash associated with Cetuximab (Erbitux®) when compared to receiving standard care for the treatment of skin rash.

DETAILED DESCRIPTION:
Of the 100 subjects who will participate in this study, 50 will be in the extensive treatment group and 50 will be in the standard care group. Subjects in the extensive treatment group will use Doxycycline capsule, 100 mg, taken twice daily, sunscreen SPF 30 or higher, moisturizer applied to the face, hands, feet, neck, back, and chest each morning after sunscreen, hydrocortisone 1% cream applied to the face, hands, feet, neck, back, and chest each evening.

Subjects will start taking the capsule and applying the creams three days prior to beginning cetuximab therapy. They will continue this regimen of taking the capsule and applying the creams for 8 weeks. If they develop severe skin rash as a result of cetuximab therapy, the study doctor may decide to reduce the amount of the dose of cetuximab that they receive or prescribe other medicines according to standard treatment recommendations, just as he/she would if the subject was not participating in this study. Subjects will be monitored at enrollment, 3 weeks into cetuximab treatment and at the end of cetuximab treatment for adherence, side effects and quality of life.

The standard care group will not receive preventive treatment, but they will be allowed to use sunscreen and moisturizer if desired. They, too, will be monitored at enrollment, 3 weeks into cetuximab treatment and at the end of cetuximab treatment for adherence, side effects and quality of life.

If a subject is assigned to this group and they develop a severe skin rash, the study doctor will treat their rash according to standard treatment recommendations, which may include Hydrocortisone 1% cream, Doxycycline capsules or other medications.

There will be a follow-Up period for both extensive treatment and standard care groups. At 6 months, 12 months, 18 months and 24 months, after the end of the subject's 8 week study treatment period, they will be contacted by telephone or discussed during their routine clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Diagnosis of colorectal or head and neck cancer
3. Receipt of at least one dose of cetuximab during the study time period

Exclusion Criteria:

1. Prior cetuximab treatment within the 6 months of study initiation
2. Current treatment with tyrosine kinase inhibitors
3. Patients who are pregnant or incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Rash | Change from Baseline, week 3, week 8
  Evaluate the incidence of cetuximab-induced rash, Compare the severity of cetuximab-induced rash between the extensive treatment group (ETG) and the standard care group (SCG).

SECONDARY OUTCOMES:
Quality of Life (QOL) | Change from Baseline, week 3, week 8
  Estimate and compare the quality of life (QOL) between the extensive treatment group and standard treatment group.
Adherence to treatment regimen | Change in adherence from baseline to week 8
  Estimate and compare adherence rate in Extensive Treatment Group and Standard Treatment Group
Progression Free Survival | Surival Follow up (6 months, 12 months, 18 months, and 24 months)
  Estimate and compare Progression-Free Survival (PFS) in extensive treatment group and standard treatment group. Survival follow-ups will be at 6 months, 12 months, 18 months, and 24 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A. Redman, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States